CLINICAL TRIAL: NCT05343143
Title: An Open-Label, Multicenter, Pilot Study to Evaluate the Performance and Safety of NeuraGen® 3D Nerve Guide Matrix.
Brief Title: NeuraGen 3D Pilot Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow Enrollment, Sponsor Decision
Sponsor: Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T-NERVE3D-001
Record Dates: First submitted 2022-04-18; First posted 2022-04-25 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Digital Nerve Injury

STUDY DESIGN:
Intervention Model Description: single arm investigational clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- NeuraGen 3D Nerve Guide Matrix (Other): Integra NeuraGen 3D Nerve Guide Matrix is a resorbable implant for the repair of peripheral nerve gaps.
  Interventions: Device: NeuraGen 3D Nerve Guide Matrix

INTERVENTIONS:
Device: NeuraGen 3D Nerve Guide Matrix — Integra NeuraGen 3D Nerve Guide Matrix is a resorbable implant for the repair of peripheral nerve gaps.

SUMMARY:
This is a 10-subject, 12-month follow-up, prospective, multi-center, open-label, single arm clinical trial designed to understand the initial performance characteristics and confirm the safety profile of the NeuraGen 3D Nerve Guide Matrix.

DETAILED DESCRIPTION:
The NeuraGen® 3D Nerve Guide Matrix is indicated for the repair of peripheral nerve discontinuities where tension-free closure can be achieved by flexion of the digit or extremity.

ELIGIBILITY:
Key Inclusion Criteria:

* Subject has one, single level, digital nerve injury that:
* Involves complete traumatic nerve section of the common or proper nerve of the palmar aspect of hand.
* Occurred less than and up to 21 days prior to the nerve repair surgery detailed in this protocol.
* In the opinion of the investigator, has a gap which can be easily closed without placing undue tension on the ends of the nerves with the device (i.e., the gap must be shorter than the maximum length of the device being used).
* Subject has adequate vascular perfusion of the target hand as assessed by the investigator
* Subject can accommodate immobilization of the injured hand post-operatively.
* Subject's contralateral hand is intact and of normal function.

Exclusion Criteria:

* Nerve to be repaired is a mixed motor nerve
* Subject has a known history of hypersensitivity to bovine-derived or chondroitin-based materials.
* Subject's hand injury is of a nature which could negatively impact healing of the target nerves such as a crush or avulsion injury, incomplete transection of the target nerve, or complete separation of the digit affiliated with the target nerve.
* Subject's hand injury or general physical presentation of the target hand is of a nature which would prevent adequate measurement of functional nerve healing assessments.
* Subject has gross contamination of the wound in which the nerve to be studied in this protocol resides (i.e., presence of glass, metal, other large debris).
* Subject has pre-existing nerve lesions or known diagnosis of compressive neuropathy of median or ulnar nerves (i.e., Cubital or carpal tunnel syndrome).
* Subject has an active infection of the area around the nerve defect.
* Subject has unstable vital signs.
* Subject has a disorder known to affect the peripheral nervous system (PNS) such as:
* Subject has any systemic disease which may confound study results Subject is known to have received immunosuppressive or antineoplastic agents or systemic steroids within 7 days of the study.
* Subject is known to have had or will require radiation or other therapy to the target hand or limb which may impact nerve healing.
* Subject has a history of injury to or a congenital abnormality of the target hand or limb which may impact nerve healing or confound study results.
* Subject is pregnant (determined either by the subject's confirmation or a formal test).
* Subject has participated in another clinical trial using an investigational drug or device within 30 days prior to the nerve repair surgery detailed in this protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-05-15 (Actual); Primary Completion 2023-07-11 (Actual); Study Completion 2024-05-13 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to evaluate return to sensory recovery with the NeuraGen 3D Nerve Guide Matrix in a small group of subjects with primary nerve injury of the hand.(s2PD) at each post-operative timepoint of the study. | 12 Months
  To be assessed during in office visits using the DeMayo 2-point discrimination device

SECONDARY OUTCOMES:
Moving 2 Point Discrimination Test (m2PD) at each post-operative timepoint of the study: | 12 Months
  To be assessed during in office visits using the DeMayo 2-point discrimination device
Grip Strength Test at each post-operative timepoint of the study | 12 Months
  To be assessed during in office visits using the Camry hand dynamometer
Pinch Strength Test at each post-operative timepoint of the study | 12 Months
  To be assessed during in office visits using the Baseline Digital Pinch Gauge
Semmes-Weinstein Monofilament Testing at each post-operative timepoint of the study | 12 Months
  To be assessed during in office visits using the Baseline Tactile Semmes-Weinstein monofilament
Disabilities of the Arm, Shoulder and Hand (DASH) Score at each post-operative timepoint of the study | 12 Months
  To be completed via in office visits
Michigan Hand Outcomes Questionnaire (MHQ) at each post-operative timepoint of the study | 12 Months
  To be completed via in office visits
Continuous Visual Analog Scale for Pain at each post-operative timepoint of the study | 12 Months
  0-100 Scale, 0-no pain at all, 100- worst possible pain. To be completed via in office visits

CONTACTS AND LOCATIONS:
Overall Officials: Maria Leonard, Study Director — Integra LifeSciences
Locations (4):
- United States (4):
  - Hospital for Special Surgery, New York, New York
  - Duke University, Durham, North Carolina
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania